CLINICAL TRIAL: NCT04348682
Title: Expanded Access Protocol of 68Ga-PSMA-11 for Prostate Cancer PET Imaging
Brief Title: Expanded Access Protocol of 68Ga-PSMA-11 for PET Imaging
Status: Approved for marketing | Type: Expanded Access
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 19-001868
Record Dates: First submitted 2020-03-13; First posted 2020-04-16 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Prostate Cancer
Keywords: prostate; imaging
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Positron-Emission Tomography

STUDY DESIGN:
Expanded Access Types: Individual, Intermediate

INTERVENTIONS:
Diagnostic Test: Positron Emission Tomography (PET) Imaging — A single dose activity of 5 mCi (accepted range of 3-7 mCi) of 68Ga-PSMA-11 will be intravenously administered to patient as a bolus injection. After 50-100 minutes of uptake time, the patient will undergo a whole body (skull to mid-thighs) PET/CT imaging.

SUMMARY:
To provide expanded access to 68Ga-PSMA-11 PET imaging for eligible participants to detect and localize prostate cancer for initial and subsequent treatment strategy.

DETAILED DESCRIPTION:
Prostate-specific membrane antigen (PSMA) targeted Positron Emission Tomography (PET) imaging has been embraced enthusiastically worldwide. Given the unmet clinical need for accurately diagnosing and staging prostate cancer and the encouraging results of 68Ga-PSMA-11 PET worldwide, University of California Los Angeles (UCLA) and University of California San Francisco (UCSF) conducted pivotal registration trials to assess 68Ga-PSMA-11's safety and efficacy profile in detecting prostate cancer in adult patients. To gap the unmet clinical need of 68Ga-PSMA-11 PET during the period prior to FDA approval, UCLA Nuclear Medicine offers expanded access of this investigational PET drug to eligible participants.

ELIGIBILITY:
Biochemical recurrent (i. Inclusion/Exclusion) and preprostatectomy (ii. Inclusion/Exclusion) staging patients will be eligible for the expanded access protocol. In order to be eligible to participate in this study, an individual must meet the following criteria:

Biochemical Recurrence Population:

i. Inclusion Criteria:

* Histopathological proven prostate adenocarcinoma.
* Rising prostatic specific antigen(PSA) after definitive therapy with prostatectomy or radiation therapy.

  * Post radical prostatectomy (RP)
  * PSA equals to or greater than 0.2 ng/mL measured more than 6weeks after RP
  * Post-radiation therapy -ASTRO-Phoenix consensus definition
  * Nadir + greater than or equal to 2 ng/mL rise in PSA
* Karnofsky performance status of ≥ 50 (or Eastern Cooperative Oncology Group (ECOG)/ World Health Organization (WHO) equivalent).
* Age > 18.
* Ability to understand a written informed consent document, and the willingness to sign it.

  i. Exclusion Criteria:
* Concomitant investigational therapy.
* Known inability to lie flat, remain still or tolerate a PET scan.
* Patient undergoing active treatment for non-prostate malignancy, other than skin basal cell or cutaneous superficial squamous cell carcinoma that has not metastasized and superficial bladder cancer.

Preprostatectomy Staging Population:

ii. Inclusion criteria:

* Biopsy proven prostate adenocarcinoma.
* Considered for prostatectomy with lymph node dissection.
* Intermediate to high-risk disease (as determined by elevated PSA [PSA>10], T-stage [T2b or greater], Gleason score [Gleason score > 6] or other risk factors).
* Able to provide written consent.
* Karnofsky performance status of ≥50 (or ECOG/WHO equivalent).

ii. Exclusion criteria:

* Patients not capable of getting PET study due to weight, claustrophobia, or inability to lay still for the duration of the exam.
* Neoadjuvant chemotherapy, radiation therapy or any definitive local therapy prior to prostatectomy including focal ablation techniques (HiFu).

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Participation is not based on self-representation. Participation is based on the possession of a prostate gland.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie Calais, M.D., Principal Investigator — University of California at Los Angeles
Locations (1):
- University of California at Los Angeles, Los Angeles, California, United States